CLINICAL TRIAL: NCT02983578
Title: Phase II Clinical Trial Evaluating Intravenous AZD9150 (Antisense STAT3) With MEDI4736 (Anti-PD-L1) in Patients With Advanced Pancreatic, Non-Small Cell Lung Cancer, and Mismatch Repair Deficient Colorectal Cancer
Brief Title: Danvatirsen and Durvalumab in Treating Patients With Advanced and Refractory Pancreatic, Non-Small Cell Lung Cancer, and Mismatch Repair Deficient Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0108; NCI-2018-01296 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0108 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-12-01; First posted 2016-12-06 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Advanced Colorectal Carcinoma; Advanced Lung Non-Small Cell Carcinoma; Lung Non-Small Cell Carcinoma; Mismatch Repair Deficiency; Refractory Colorectal Carcinoma; Refractory Lung Carcinoma; Refractory Pancreatic Carcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Turcot syndrome; Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms | interventions — danvatirsen; durvalumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (danvatirsen, durvalumab) (Experimental): Patients receive danvatirsen IV over 1 hour on days 7, 5 and 3 prior to cycle 1, then on days 1, 8, 15 and 22. Patients also receive durvalumab IV over 1 hour on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Danvatirsen; Biological: Durvalumab

INTERVENTIONS:
Drug: Danvatirsen — Given IV
  Other Names: AZD9150; ISIS 481464; ISIS-STAT3rx
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736

SUMMARY:
This phase II trial studies how well danvatirsen and durvalumab work in treating patients with pancreatic cancer, non-small cell lung cancer and mismatch repair deficient colorectal cancer that has spread to other places in the body and does not respond to treatment. Danvatirsen may be used to block the production of proteins needed for tumor cell growth. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving danvatirsen and durvalumab may work better at treating pancreatic cancer, non-small cell lung cancer and mismatch repair deficient colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate disease control rate (DCR) at 4 months. II. Evaluate tumor-based biomarkers in paired pre and post treatment biopsies (10 in each arm, 30 total) that may correlate with treatment or prospectively identify patients likely to respond to treatment with danvatirsen (AZD9150) in combination with durvalumab (MEDI4736) (may include PD-L1 expression, phosphorylated or total STAT3 expression, tumor genetics, characterization of immune infiltrates, or other stratification markers).

III. Explore the relationship between PD-L1 protein levels in the membrane of circulating tumor cells obtained by peripheral blood draws prior to, during, and after treatment with clinical endpoints including treatment efficacy and toxicity.

SECONDARY OBJECTIVES:

I. Evaluate the frequency of dose limiting toxicities. II. Evaluate frequency of objective response (as defined as partial response [PR] or complete response [CR] according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria).

III. Evaluate duration of response (DOR) measured from the time measurement criteria are first met for CR or PR, whichever is first recorded, until the first date that recurrent or progressive disease (PD) is objectively documented.

IV. Evaluate best overall response (including CR, PR, stable disease [SD], and PD, according to RECIST version 1.1 criteria).

V. Evaluate progression free survival (PFS) from allocation to the first documentation of PD as determined by the investigator or death from any cause, whichever occurs first.

EXPLORATORY OBJECTIVES:

I. Explore the relationship between radiologic metrics (radiomics) prior to, during, and after treatment with clinical endpoints including treatment efficacy and toxicity.

OUTLINE:

Patients receive danvatirsen intravenously (IV) over 1 hour on days 7, 5 and 3 prior to cycle 1, then on days 1, 8, 15 and 22. Patients also receive durvalumab IV over 1 hour on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 1-3 months, then every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The patient/legal representative must be able to read and understand the informed consent form (ICF) and must have been willing to give written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the United States of America [USA]; European Union Data Privacy Directive in the European Union [EU]) before any study-specific procedures, including screening evaluations, sampling, and analyses
* Has a histological confirmation of pancreatic cancer, mismatch deficient colorectal cancer, or non-small cell lung cancer (NSCLC) that is refractory to standard therapy or for which no standard of care regimen currently exists
* Has an Eastern Cooperative Oncology Group (ECOG) performance score (PS) score of 0 or 1
* Has measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) with a minimum size of 10 mm by computerized tomography (CT) scan, except lymph nodes which must have minimum short axis size of 15 mm (CT scan slice thickness no greater than 5 mm in both cases). Indicator lesions must not have been previously treated with surgery, radiation therapy, or radiofrequency ablation unless there is documented progression after therapy
* Transfusions intended to elevate any parameters below solely for the intent of meeting study eligibility are not permitted
* Leukocytes >= 3000 mcL
* Absolute neutrophil count >= 1500 mcL
* Platelets > = 100 000 mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 3 x ULN in patients with documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or in the presence of liver metastases
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN if no demonstrable liver metastases or =< 5 x ULN in the presence of liver metastases
* Creatinine within normal limits OR, for patients with levels above institutional normal: creatinine clearance measured by 24-hour urine collection >= 60 mL/min, OR calculated corrected creatinine clearance >= 60 mL/min/1.73 m^2 using the Cockcroft-Gault formula (Cockcroft and Gault 1976) corrected for the body surface area
* Women of childbearing potential and men who are sexually active with a female partner of childbearing potential must be surgically sterilized, practicing abstinence, or agree to use 2 birth control methods before study entry, for the duration of study participation, and for 20 weeks after the final dose of study drug; cessation of birth control after this point should be discussed with a responsible physician. Women of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause). Two methods of contraception which are considered accurate per protocol must be combined. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control
* Women of childbearing potential also may not be breast feeding and must have a negative serum or urine pregnancy test within 72 hours before the start of study treatment
* The patient/legal representative must be willing to provide written consent for collection of formalin fixed paraffin-embedded blocks or slides from archival diagnostic histology samples, where available

Exclusion Criteria:

* Has a spinal cord compression unless asymptomatic, radiographically stable over the last 4 weeks, and not requiring steroids for at least 4 weeks before the start of study treatment
* Presently has a second malignancy other than squamous cell carcinoma of the head and neck (SCCHN), or history of treatment for invasive cancer other than SCCHN in the past 3 years. Exceptions are:

  * Previously treated in-situ carcinoma (i.e., noninvasive)
  * Cervical carcinoma stage 1B or less
  * Noninvasive basal cell and squamous cell skin carcinoma
  * Radically treated prostate cancer (prostatectomy or radiotherapy) with normal prostate-specific antigen, and not requiring ongoing antiandrogen hormonal therapy
* Patients must have completed previous cancer-related treatments before enrollment. Any concurrent chemotherapy, radiotherapy, immunotherapy, or biologic, or hormonal therapy for cancer excludes the patient (concurrent use of hormones for noncancer-related conditions [e.g., insulin for diabetes or hormone replacement therapy] is acceptable). The following intervals between end of the prior treatment and first dose of study drug must be observed:

  * Port-a-cath placement: no waiting required
  * Minor surgical procedures: >= 7 postoperative days
  * Major surgery: >= 4 weeks
  * Radiotherapy: >= 4 weeks
  * Chemotherapy: >= 4 weeks
  * Immunotherapy or investigational anticancer therapy with agents other than monoclonal antibodies (mAbs): >= 4 weeks
  * Immunotherapy or investigational anticancer therapy with mAbs: >= 6 weeks
  * Immunosuppressive medication: >= 4 weeks with the exceptions of intranasal or inhaled corticosteroids or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
* Is still experiencing toxicity related to prior treatment and assessed as Common Terminology Criteria for Adverse Events (CTCAE) grade > 1. Exceptions are alopecia and/or anorexia. The eligibility of patients who are still experiencing irreversible toxicity that is not reasonably expected to be exacerbated by the study drugs in this study (e.g., hearing loss) must be reviewed and approved by both the principal investigator and medical monitor
* Has experienced immune-related adverse events (AEs) (irAEs) while receiving prior immunotherapy (including anti-CTLA4 treatment) and assessed as CTCAE grade >= 3
* Has active or prior documented autoimmune disease within the past 2 years with the exceptions of vitiligo, Grave's disease, and/or psoriasis not requiring systemic treatment
* Has active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Has a history of primary immunodeficiency
* Has undergone an organ transplant that requires use of immunosuppressive treatment
* Has a history of interstitial lung disease or pneumonitis from any cause
* Has a history of allergic reactions attributed to the study treatments (AZD9150 or MEDI4736), their compounds, or agents of similar chemical or biologic composition (e.g., antibody therapeutics)
* Suffers from a comorbidity that in the opinion of the investigator renders the patient unsuitable for participation in the study. Such comorbidity may include, but is not limited to, uncontrolled intercurrent illness such as active infection, severe active peptic ulcer disease or gastritis, myocardial infarction within 6 months before entry, congestive heart failure, symptomatic congestive heart failure, active cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* As judged by the investigator, has any evidence of severe or uncontrolled systemic diseases such as active bleeding diatheses, is positive for human immunodeficiency virus (HIV), or has active hepatitis B virus (HBV) and/or hepatitis C virus (HCV)
* Has a known history of tuberculosis
* Has a condition that, in the opinion of the investigator, would interfere with the evaluation of the study drugs or the interpretation of patient safety or study results
* Has received a live attenuated vaccine within 28 days before the first dose of study drug
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements
* Patients with clinically active brain metastases (known or suspected) are excluded unless the brain metastases have been previously treated and are considered stable. Stable brain metastases are defined as no change on CT scan or magnetic resonance imaging (MRI) scan for a minimum of 2 months AND no change in steroid dose for a minimum of 4 weeks, unless change due to intercurrent infection or other acute event
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), serious AEs | Up to 4 years
Physiological parameters (Laboratory evaluations) | Up to 4 years
  Blood samples for routine coagulation assessments will be obtained at screening and once during week 4 of cycle 1.
Incidence of treatment-emergent AEs (TEAEs), SAEs and death(s) | Up to 4 years
  Will be graded in accordance with National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03.
PD-L1 expression | Up to 4 years
Phosphorylated or total STAT3 expression levels | Up to 4 years
Characterization of immune infiltrates | Up to 4 years
Quantification and characterization of CD8 staining pattern | Up to 4 years
PD-L1 protein levels in the membrane of circulating tumor cells | Baseline up to 4 years
Physiological parameters | Up to 4 years
  Vital signs will required at screening before dosing on Day -7 of the Lead-in; before dosing on Days 1, 8, 15, and 22 of each cycle; and at the EOT visit.
Physical Examinations | Up to 4 years
  A complete physical examination is required at screening, before dosing on Day 7 of the Lead in, before dosing on Day 1 of each cycle, and at the EOT visit. A targeted physical examination as directed by disease, signs and symptoms is required before dosing on Day 15 of each cycle.

SECONDARY OUTCOMES:
Disease control | At 4 months
  Will be defined as a compete response (CR), partial response (PR) or stable disease (SD), according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
Objective response | Up to 4 years
  Will be defined as a CR or PR according to RECIST version 1.1.
Duration of response according to RECIST version 1.1 criteria | From the time measurement criteria are first met for CR or PR, assessed up to 4 years
Best overall response (including CR, PR, SD, and progressive disease [PD], according to RECIST version 1.1 criteria) | Up to 4 years
Progression free survival | From allocation assessed up to 4 years
Overall survival | From start of treatment assessed up to 4 years

OTHER OUTCOMES:
Radiomic measurements | Baseline up to 4 years
  These are IRECIST measurements

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Tang C, Hartley GP, Couillault C, Yuan Y, Lin H, Nicholas C, Srinivasamani A, Dai J, Dumbrava EEI, Fu S, Karp DD, Naing A, Piha-Paul SA, Rodon Ahnert J, Pant S, Subbiah V, Yap TA, Tsimberidou AM, Guerrero P, Dhebat S, Proia T, Curran MA, Hong DS. Preclinical study and parallel phase II trial evaluating antisense STAT3 oligonucleotide and checkpoint blockade for advanced pancreatic, non-small cell lung cancer and mismatch repair-deficient colorectal cancer. BMJ Oncol. 2024 Jul 30;3(1):e000133. doi: 10.1136/bmjonc-2023-000133. eCollection 2024. PMID 39886125
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org